CLINICAL TRIAL: NCT01208935
Title: Safety, Tolerability and Efficacy of the Nicotine Patch and Gum for the Treatment of Adolescent Tobacco Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Steve Heishman, NIDA IRP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-IRP-322
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-09

CONDITIONS: Tobacco Dependence
Keywords: Randomized; Double blind; double-dummy; placebo-controlled
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Nicotine Patch
Drug: Nicotine Gum

SUMMARY:
The purpose of this study is to test the safety, tolerability, compliance and efficacy of two different forms of nicotine replacement therapy (NRT) (the nicotine transdermal patch and the nicotine gum) in a nicotine-dependent adolescent population.

DETAILED DESCRIPTION:
We hypothesize that two nicotine replacement delivery systems (patch and gum) are both safe and efficacious for the treatment of adolescent nicotine dependence. Consequently, use of both the patch and gum should be tolerable in this population with only minor adverse side-effects. Secondly, some individuals in both groups (patch, gum) may benefit from either cessation or reduction in smoke exposure, as a result of the distinctly different mechanisms of the two treatments (steady state vs. intermittent delivery of NRT).

A.The primary objectives of this study are:

1. to evaluate the comparative safety of the nicotine transdermal system (21 mg "patch") and the nicotine gum (2 mg and 4 mg), dosed appropriately to pre-treatment levels of smoking, to initiate and sustain smoking cessation and reduction ;
2. to compare compliance levels with the patch and gum;
3. to evaluate the comparative efficacy of the patch and the gum to initiate and sustain smoking cessation and reduction;
4. to compare the rates of biochemically-verified continuous abstinence by using intent-to-treat analysis based on individual subject outcome.

B.The secondary objectives of this study are:

1. to correlate pre-treatment nicotine exposure (saliva cotinine) with withdrawal intensity measured in all groups during treatment and with treatment outcome;
2. to compare biological markers of smoke exposure (expired air CO and saliva thiocyanate) with self-reports of smoking and to correlate them with withdrawal symptomatology and treatment outcome;
3. to obtain smoking topography data (puff volume, velocity of intake, interpuff interval, and puffs per cigarette) on adolescent patterns of smoking as an index of smoking intensity and exposure and to correlate pre-treatment smoking intensity with treatment outcome.

C.The tertiary objectives are:

1. to examine the validity of the use of biochemical markers of smoke exposure (expired air CO and saliva thiocyanate) as potential markers of smoking cessation in adolescents;
2. to compare the relative cotinine exposure of adolescents who are smoking with those who are receiving nicotine replacement who do and do not successfully quit

ELIGIBILITY:
Inclusion Criteria:

* History of smoking 11 or more cigarettes per day (cpd) for at least one year
* Fagerström Test for Nicotine Dependence score of 5 and above
* General good health as verified by history, physical, psychiatric examination and screening laboratory tests

Exclusion Criteria:

* History of cardiac disease
* Active dependence on any drug other than nicotine (as assessed by the DUSI)
* Current or past severe psychiatric disorders as per the Diagnostic Interview for Children and Adolescents (DICA-A)
* Current use of tobacco or nicotine containing products other than cigarettes
* Previous use of any nicotine transdermal patch or nicotine gum
* Presence or history of severe skin allergies or dermatoses
* Pregnancy or lactation
* Active oral, dental or jaw mobility problems

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 1999-08; Primary Completion 2004-06 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
a)Safety will be tabulated as a function of reported and observed adverse side-effects.
b)Tolerability and Compliance by attendance at visits, completeness of smoking cessation diaries, saliva cotinine, and correlations of biologic markers (expired air CO and saliva thiocyanate) with smoking cessation diaries.
c) Efficacy by Minnesota Withdrawal scale, craving visual analog scales and Questionnaire of Smoking Urges, smoking abstinence/reduction (as per self-reported data in smoking cessation diaries), expired air CO and saliva thiocyanate.
d) Weight and body mass index (BMI)
e)Cognitive performance tests

CONTACTS AND LOCATIONS:
Overall Officials: Eric T. Moolchan, M.D., Principal Investigator — National Institutes on Drug Abuse IRP/ NIH
Locations (1):
- Teen Tobacco Addiction Research Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Background] Moolchan ET, Robinson ML, Ernst M, Cadet JL, Pickworth WB, Heishman SJ, Schroeder JR. Safety and efficacy of the nicotine patch and gum for the treatment of adolescent tobacco addiction. Pediatrics. 2005 Apr;115(4):e407-14. doi: 10.1542/peds.2004-1894. PMID 15805342
- [Background] Aung AT, Pickworth WB, Moolchan ET. History of marijuana use and tobacco smoking topography in tobacco-dependent adolescents. Addict Behav. 2004 Jun;29(4):699-706. doi: 10.1016/j.addbeh.2004.02.012. PMID 15135551
- [Background] Zimmerman DM, Sehnert SS, Epstein DH, Pickworth WB, Robinson ML, Moolchan ET. Smoking topography and trajectory of asthmatic adolescents requesting cessation treatment. Prev Med. 2004 Nov;39(5):940-2. doi: 10.1016/j.ypmed.2004.03.032. PMID 15475027
- [Background] Moolchan ET, Zimmerman D, Sehnert SS, Zimmerman D, Huestis MA, Epstein DH. Recent marijuana blunt smoking impacts carbon monoxide as a measure of adolescent tobacco abstinence. Subst Use Misuse. 2005;40(2):231-40. doi: 10.1081/ja-200048461. PMID 15770886
- [Background] Moolchan ET, Hudson DL, Schroeder JR, Sehnert SS. Heart rate and blood pressure responses to tobacco smoking among African-American adolescents. J Natl Med Assoc. 2004 Jun;96(6):767-71. PMID 15233486
- [Background] Jones DN, Schroeder JR, Moolchan ET. Time spent with friends who smoke and quit attempts among teen smokers. Addict Behav. 2004 Jun;29(4):723-9. doi: 10.1016/j.addbeh.2004.02.026. PMID 15135554
- [Background] Cramer K, Tuokko HA, Mateer CA, Hultsch DF. Measuring awareness of financial skills: reliability and validity of a new measure. Aging Ment Health. 2004 Mar;8(2):161-71. doi: 10.1080/13607860410001649581. PMID 14982721
- [Background] Moolchan ET, Schroeder JR. Quit attempts among African American teenage smokers seeking treatment: gender differences. Prev Med. 2004 Dec;39(6):1180-6. doi: 10.1016/j.ypmed.2004.04.050. PMID 15539053
- [Background] Robinson ML, Berlin I, Moolchan ET. Tobacco smoking trajectory and associated ethnic differences among adolescent smokers seeking cessation treatment. J Adolesc Health. 2004 Sep;35(3):217-24. doi: 10.1016/j.jadohealth.2003.10.005. PMID 15313503
- [Background] Aung AT, Hickman NJ 3rd, Moolchan ET. Health and performance related reasons for wanting to quit: gender differences among teen smokers. Subst Use Misuse. 2003 Jun;38(8):1095-107. doi: 10.1081/ja-120017652. PMID 12901450
- [Background] Moolchan ET, Berlin I, Robinson ML, Cadet JL. Characteristics of African American teenage smokers who request cessation treatment: implications for addressing health disparities. Arch Pediatr Adolesc Med. 2003 Jun;157(6):533-8. doi: 10.1001/archpedi.157.6.533. PMID 12796232
- [Background] Moolchan ET, Mermelstein R. Research on tobacco use among teenagers: ethical challenges. J Adolesc Health. 2002 Jun;30(6):409-17. doi: 10.1016/s1054-139x(02)00365-8. PMID 12039510
- [Background] Moolchan ET, Berlin I, Robinson ML, Cadet JL. African-American teen smokers: issues to consider for cessation treatment. J Natl Med Assoc. 2000 Dec;92(12):558-62. PMID 11202758
- [Background] Moolchan ET, Ernst M, Henningfield JE. A review of tobacco smoking in adolescents: treatment implications. J Am Acad Child Adolesc Psychiatry. 2000 Jun;39(6):682-93. doi: 10.1097/00004583-200006000-00006. PMID 10846302
- [Background] Collins CC, Moolchan ET. Shorter time to first cigarette of the day in menthol adolescent cigarette smokers. Addict Behav. 2006 Aug;31(8):1460-4. doi: 10.1016/j.addbeh.2005.10.001. Epub 2005 Nov 21. PMID 16303257
- [Background] Franken FH, Pickworth WB, Epstein DH, Moolchan ET. Smoking rates and topography predict adolescent smoking cessation following treatment with nicotine replacement therapy. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):154-7. doi: 10.1158/1055-9965.EPI-05-0167. PMID 16434603
- [Background] Robinson ML, Schroeder JR, Moolchan ET. Adolescent smokers screened for a nicotine replacement treatment trial: correlates of eligibility and enrollment. Nicotine Tob Res. 2006 Jun;8(3):447-54. doi: 10.1080/14622200600670413. PMID 16801302
- [Background] Moolchan ET, Franken FH, Jaszyna-Gasior M. Adolescent nicotine metabolism: ethnoracial differences among dependent smokers. Ethn Dis. 2006 Winter;16(1):239-43. PMID 16599377
- [Background] Moolchan ET, Aung AT, Henningfield JE. Treatment of adolescent tobacco smokers: issues and opportunities for exposure reduction approaches. Drug Alcohol Depend. 2003 Jun 5;70(3):223-32. doi: 10.1016/s0376-8716(03)00012-7. PMID 12757960